CLINICAL TRIAL: NCT06777589
Title: Exploration of the Range of the Quantitative Nociception Index (qNOX) During Gastrointestinal Endoscopy Under Intravenous Sedation: a Multicenter Clinical Study
Brief Title: Quantitative Consciousness Index Monitoring (qNOX) of Sedation During Endoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Min Su (Other)
Responsible Party: Sponsor-Investigator, Min Su, Professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202410901
Record Dates: First submitted 2025-01-02; First posted 2025-01-16 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Nociception
Keywords: Nociception; endoscopy; Depth of anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group Ⅰ: Propofol Gastroscopy Group (GP Group) (Experimental): During the gastroscopy procedure, the Bispectral Index Monitor (Apollo-9000A) was utilized to monitor patients' qCON and qNOX. The anesthesia sedation protocol involved induction with propofol, with an induction dose ranging from 1.5 to 2.5 mg/kg. The propofol was administered using a syringe pump at an infusion rate of 300 ml/h. During the examination, propofol was infused at a rate of 4 to 6 mg/kg·h.
  Interventions: Device: Monitoring of anesthesia depth
- Group Ⅱ: Propofol Combined with Low-dose Sufentanil Gastroscopy Group (GSP Group) (Experimental): During the gastroscopy procedure, the Bispectral Index Monitor (Apollo-9000A) was used to monitor patients' qCON and qNOX. The anesthesia sedation protocol involved induction with a combination of propofol and a low dose of sufentanil. Initially, sufentanil 5μg (1μg/mL) was administered intravenously, followed by the initiation of propofol infusion one minute later using a syringe pump. The induction dose of propofol was 1.5 to 2.5 mg/kg, with a propofol infusion rate of 300 ml/h. During the examination, propofol was infused at a rate of 4 to 6 mg/kg·h.
  Interventions: Device: Monitoring of anesthesia depth
- Group Ⅲ: Propofol Colonoscopy Group (CP Group) (Experimental): During the Colonoscopy procedure, the Bispectral Index Monitor (Apollo-9000A) was utilized to monitor patients' qCON and qNOX. The anesthesia sedation protocol involved induction with propofol, with an induction dose ranging from 1.5 to 2.5 mg/kg. The propofol was administered using a syringe pump at an infusion rate of 300 ml/h. During the examination, propofol was infused at a rate of 4 to 6 mg/kg·h.
  Interventions: Device: Monitoring of anesthesia depth
- Group IV: Propofol Combined with Low-dose Sufentanil Colonoscopy Group (CSP Group) (Experimental): During the Colonoscopy procedure, the Bispectral Index Monitor (Apollo-9000A) was used to monitor patients' qCON and qNOX. The anesthesia sedation protocol involved induction with a combination of propofol and a low dose of sufentanil. Initially, sufentanil 5μg (1μg/mL) was administered intravenously, followed by the initiation of propofol infusion one minute later using a syringe pump. The induction dose of propofol was 1.5 to 2.5 mg/kg, with a propofol infusion rate of 300 ml/h. During the examination, propofol was infused at a rate of 4 to 6 mg/kg·h.
  Interventions: Device: Monitoring of anesthesia depth

INTERVENTIONS:
Device: Monitoring of anesthesia depth — During gastroscopy and colonoscopy procedures, the Bispectral Index Monitor (Apollo-9000A) is utilized to monitor patients' quantitative consciousness index (qCON) and quantitative nociception index (qNOX).

SUMMARY:
Nociception is the encoding and processing of noxious stimulation and is considered an objective indicator for monitoring pain. Currently, a new clinically-applied medical-engineering integrated monitoring device for noxious stimulation response has emerged. Its fundamental principle is based on the monitoring of electroencephalographic (EEG) activity, incorporating two monitoring parameters: the quantitative consciousness (qCON) index and the quantitative nociceptive (qNOX) index. This device enables more precise monitoring of anesthesia depth, quantification of patients' anesthesia analgesia and stress levels, and reliable monitoring of responses to noxious stimulation. During tracheal intubation for general anesthesia, when the qCON value falls within the range of 40 to 60 and the qNOX value is between 30 and 50, it indicates that the patient is in an appropriate state of sedation and analgesia. However, there is currently no universally acknowledged standard for the optimal qNOX reference range during conscious sedation endoscopy. Therefore, this study utilizes the noxious stimulation response index (qNOX) to monitor noxious stimulation during the procedure, aiming to identify the best timing for inserting the endoscope during conscious sedation endoscopy and explore the appropriate range of qNOX for this purpose.

DETAILED DESCRIPTION:
This is a multicenter clinical study. Study Objective: To explore the reasonable range of the qNOX and the optimal timing for gastroscopy and colonoscopy during intravenous sedation-assisted endoscopic examinations. Study Protocol: A total of 900 patients undergoing intravenous sedation-assisted digestive endoscopy in the outpatient clinics of the participating institutions were selected. Among them, 450 patients undergoing gastroscopy were divided into a propofol group (GP group) and a propofol combined with low-dose sufentanil group (GSP group); 450 patients undergoing colonoscopy were divided into a propofol group (CP group) and a propofol combined with low-dose sufentanil group (CSP group). The bispectral index monitor (Apollo-9000A) was used to monitor the qCON and qNOX of patients during intravenous sedation-assisted digestive endoscopy. The values of qCON, qNOX, SBP (systolic blood pressure), DBP (diastolic blood pressure), MAP (mean arterial pressure), HR (heart rate), SpO2 (peripheral capillary oxygen saturation), and MOAA/S (Modified Observer's Assessment of Alertness/Sedation) scores at different time points during gastroscopy and colonoscopy were observed and recorded. The occurrence of adverse events during and after the examinations was also documented.

ELIGIBILITY:
Inclusion Criteria

1. Age between 18 and 60 years old;
2. ASA-PS (American Society of Anesthesiologists Physical Status) classification of I to II;
3. Body Mass Index (BMI): 18 to 28 kg/m²;
4. Patients undergoing diagnostic and therapeutic procedures under sedation for lower gastrointestinal endoscopy;
5. Clear understanding and voluntary participation in this study, with informed consent signed.

Exclusion Criteria

1. Patients requiring complex endoscopic techniques for diagnosis and treatment;
2. Patients who have participated in other clinical trials in the past three months;
3. Pregnant and lactating patients;
4. Patients with allergies to sedatives/anesthetics and other severe anesthesia risks;
5. Patients with preoperative chronic pain or a history of substance abuse;
6. Patients with severe neurological diseases such as stroke, hemiplegia, convulsions, epilepsy, etc.;
7. Patients with known difficult airways such as limited mouth opening, restricted neck and jaw movement, rheumatoid spondylitis, temporomandibular joint arthritis, etc.;
8. Patients with potentially life-threatening circulatory and respiratory diseases that are not adequately controlled, such as uncontrolled severe hypertension, severe arrhythmias, unstable angina pectoris, acute respiratory infections, asthma exacerbations, etc.;
9. Patients with liver dysfunction (Child-Pugh Class C or higher), acute upper gastrointestinal bleeding with shock, severe anemia, gastrointestinal obstruction with gastric retention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The value of qNOX | Start of the procedure，when the gastroscope passes through the pharynx or the colonoscope passes through the anus.
  The value of qNOX when the gastroscope passes through the pharynx or the colonoscope passes through the anus.

SECONDARY OUTCOMES:
The values of qCON 、 qNOX at different time | Up to 1 hours, from the moment the patient enters the endoscopy procedure room until they exit it
  The Values of qCON 、 qNOX at different time points during gastroscopy and enteroscopy ① Time points for gastroscopy: Baseline value (T0), Loss of consciousness (T1), Before insertion of the gastroscope (T2), Passage of the gastroscope through the pharynx (T3), After insertion of the gastroscope (T4), Examination completion (T5), Awakening (T6), Discharge from recovery room (T7).
  ② Time points for colonoscopy: Baseline value (T0), Loss of consciousness (T1), Before insertion of the colonoscope (T2), After insertion of the colonoscope into the anus (T3), Descending colon (T4), Splenic flexure (T5), Hepatic flexure (T6), Examination completion (T7), Awakening (T8), Discharge from recovery room (T9).
The values of qCON 、 qNOX under special events | Up to 1 hours, from the moment the patient enters the endoscopy procedure room until they exit it
  The values of qCON, qNOX score during coughing, body movement, biopsy, and polypectomy that occurred during the examination.
The values of SBP、DBP、 MAP at different time | Up to 1 hours, from the moment the patient enters the endoscopy procedure room until they exit it
  The Values of SBP、DBP、 MAP at different time points during gastroscopy and enteroscopy ① Time points for gastroscopy: Baseline value (T0), Loss of consciousness (T1), Before insertion of the gastroscope (T2), Passage of the gastroscope through the pharynx (T3), After insertion of the gastroscope (T4), Examination completion (T5), Awakening (T6), Discharge from recovery room (T7).
  ② Time points for colonoscopy: Baseline value (T0), Loss of consciousness (T1), Before insertion of the colonoscope (T2), After insertion of the colonoscope into the anus (T3), Descending colon (T4), Splenic flexure (T5), Hepatic flexure (T6), Examination completion (T7), Awakening (T8), Discharge from recovery room (T9).
The values of SBP、DBP、 MAP under special events | Up to 1 hours, from the moment the patient enters the endoscopy procedure room until they exit it
  The values of SBP、DBP、 MAP during coughing, body movement, biopsy, and polypectomy that occurred during the examination.
The values of HR at different time | Up to 1 hours, from the moment the patient enters the endoscopy procedure room until they exit it
  The Values of HR at different time points during gastroscopy and enteroscopy ① Time points for gastroscopy: Baseline value (T0), Loss of consciousness (T1), Before insertion of the gastroscope (T2), Passage of the gastroscope through the pharynx (T3), After insertion of the gastroscope (T4), Examination completion (T5), Awakening (T6), Discharge from recovery room (T7).
  ② Time points for colonoscopy: Baseline value (T0), Loss of consciousness (T1), Before insertion of the colonoscope (T2), After insertion of the colonoscope into the anus (T3), Descending colon (T4), Splenic flexure (T5), Hepatic flexure (T6), Examination completion (T7), Awakening (T8), Discharge from recovery room (T9).
The values of HR under special events | Up to 1 hours, from the moment the patient enters the endoscopy procedure room until they exit it
  The values of HR during coughing, body movement, biopsy, and polypectomy that occurred during the examination.
The values of MOAA/S at different time | Up to 1 hours, from the moment the patient enters the endoscopy procedure room until they exit it
  The Values of MOAA/S at different time points during gastroscopy and enteroscopy ① Time points for gastroscopy: Baseline value (T0), Loss of consciousness (T1), Before insertion of the gastroscope (T2), Passage of the gastroscope through the pharynx (T3), After insertion of the gastroscope (T4), Examination completion (T5), Awakening (T6), Discharge from recovery room (T7).
  ② Time points for colonoscopy: Baseline value (T0), Loss of consciousness (T1), Before insertion of the colonoscope (T2), After insertion of the colonoscope into the anus (T3), Descending colon (T4), Splenic flexure (T5), Hepatic flexure (T6), Examination completion (T7), Awakening (T8), Discharge from recovery room (T9).
The values of MOAA/S under special events | Up to 1 hours, from the moment the patient enters the endoscopy procedure room until they exit it
  The values of HR during coughing, body movement, biopsy, and polypectomy that occurred during the examination.
Adverse events | Up to 1 hours, from the moment the patient enters the endoscopy procedure room until they exit it
  Adverse events during gastroscopy and enteroscopy were recorded, including hypotension, hypertension, tachycardia, bradycardia, respiratory depression, hypoxemia, cough, body movement, nausea, vomiting, hiccup, injection pain, abdominal pain, abdominal distension, reflux aspiration.
Adverse events and complications after examination | 24 hours after procedure
  Bleeding, dizziness, blurred vision, nausea, vomiting, abdominal pain, abdominal distension were followed up 24h after the examination

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- China,Chongqing The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China